CLINICAL TRIAL: NCT00423709
Title: A Study of Allogeneic Blood Stem Cell Transplantation With Purine Analog-Based Conditioning For Patients With Advanced Hodgkin's Disease
Brief Title: Allogeneic Blood Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM97-259
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Hodgkin's Disease
Keywords: Hodgkin's Disease; Allogeneic Blood Stem Cell Transplantation; Bone Marrow Transplantation; Fludarabine; Melphalan
MeSH Terms: conditions — Hodgkin Disease | interventions — fludarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Allogeneic Blood Stem Cell Transplantation
Drug: Fludarabine
Drug: Melphalan

SUMMARY:
1. To determine the feasibility and toxicity of employing allogeneic peripheral blood stem cell transplantation after intensive but non-myeloablative chemotherapy in patients with relapsed Hodgkin's disease (HD).
2. To determine the engraftment kinetics and degree of chimerism that can be achieved with this strategy.
3. To assess the antitumor activity of this approach in high-risk HD patients and the possible presence of a graft-vs-HD effect.

DETAILED DESCRIPTION:
All patients in this study must have a plastic tube (catheter) inserted into a vein under the collarbone. Drugs and stem cells will be given through this tube.

Fludarabine will be given through the catheter once a day for four days. Patients will also receive melphalan for two days through the catheter. Patients receiving a transplant from a matched unrelated donor (i.e. not a blood relative) or a mismatched related donor (i.e. a blood relative, but not a full match) will also receive antithymocyte globulin (ATG) once a day for three days. ATG can help preventing graft-versus-host disease. All patients are expected to need blood transfusions as part of this treatment.

Beginning two days before the transplant, tacrolimus will be given through the catheter. It will be given 24 hours a day until the patient can swallow. The patient will then swallow one or more tacrolimus pills a day for about 6 months.

On the transplant day ("day 0"), the stem cells or bone marrow obtained from the donor will be infused through the catheter ("transplant"). Drugs will be given to reduce the chance of allergic reactions. Starting on day 7 after the transplant, filgrastim will be given through a needle to increase the growth of white blood cells. Methotrexate will be given by IV on days 1,3,6, 11 after the transplant. The patient may require blood transfusions for the following 2-4 weeks and sometimes longer.

Patients with progressive ("growing") Hodgkin's disease after the transplant will initially be taken off their immunosuppressive medications (tacrolimus, corticosteroids). If there is no response to this maneuver, they will be considered for infusion of additional cells from their donors, with or without preceding chemotherapy Both these maneuvers may produce a response ("shrinkage") of the tumor. Patients with persistent but stable (not "growing") disease may also be treated in a similar fashion. Potential side effects of the infusion of additional cells include graft-versus-host disease and /or a generalized drop in the blood counts. Both of these conditions can be serious or life-threatening.

Blood, urine, bone marrow and x-ray examinations will be performed as necessary to monitor the results of bone marrow transplantation. Patients may require blood and platelet transfusions. Blood tests will be done daily while hospitalized and several times a week until the blood counts recover. Bone marrow aspiration and biopsies will be performed prior to the transplant, when the donated cells show signs of engraftment, and at other times during the next 1 to 3 years to evaluate the growth of the transplant marrow, to evaluate possible recurrence of malignancy and recovery of immunity.

This is an investigational study. Up to 50 patients will be treated on this study. If the initial results are discouraging, the study may be stopped after a minimum of four patients have been enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients <65 years of age with histologically confirmed primary refractory or relapsed Hodgkin's disease. In the event of transplants from unrelated donors, the upper age limit will be 55 years.
2. Patients who failed or relapsed after an autologous transplant are eligible.
3. Patients should have responsive or stable disease on salvage chemotherapy. Patients with untreated, smoldering (i.e. not rapidly progressive) relapses are eligible. Patients who failed or relapsed after an autologous transplant are eligible.
4. Patients must have a serum bilirubin <2.0 mg/dl, serum creatinine <2.0 mg/dl, no symptomatic cardiac or pulmonary disease and a PS<2. Life expectancy not severely limited by concomitant illness (>12 weeks). Left ventricular ejection fraction >50%.
5. Patients must have an HLA-compatible donor (one-antigen mismatched related donors are acceptable) willing to donate marrow or rhG-CSF-mobilized peripheral blood stem cells . In the event of transplants from unrelated donors, only fully serologically A-, B- and DR-matched donors (including donors having a single micromismatch by DR/DQ molecular typing) will be acceptable. HLA-compatible cord blood unit will also be acceptable for recipient with a body weight of 50 kg or less.

Exclusion Criteria:

1. Patients with documented disease progression on salvage chemotherapy are not eligible.
2. Uncontrolled arrhythmia or symptomatic cardiac disease. FEV1, FVC and DLCO less than 50% . Symptomatic pulmonary disease. Evidence of chronic active hepatitis or cirrhosis.
3. Active or uncontrolled infection.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1998-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Anderlini, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org